CLINICAL TRIAL: NCT06942689
Title: Determination of the Optimal Volume of Liposomal Bupivacaine in Single-Shot Adductor Canal Block for Knee Joint Surgery-A Phase I/II Trial
Brief Title: Determination of the Optimal Volume of Liposomal Bupivacaine in Adductor Canal Block for Knee Joint Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hongwei Shi, Director, Department of Anesthesia, Pain and Perioperative Medicine, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20250327-13
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Optimal Volume of Liposomal Bupivacaine
Keywords: Liposomal Bupivacaine; Adductor Canal Block; Knee Surgery; Maximum Tolerated Volume; Quadriceps Muscle Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adductor Canal Block (Experimental): Phase I: The Bayesian Optimal Interval (BOIN) design is adopted to evaluate the volume escalation of liposomal bupivacaine (10, 15, 20, 25, 30, 35, 40 mL). There are 3 cases in each group, with an initial volume of 20 mL (referring to previous ACB studies d). The target incidence of adverse events (quadriceps femoris muscle strength decline ≥ 25%) is set at 10%, and the maximum volume is limited to 40 mL to avoid local anesthetic toxicity.
  Phase II: Cohort expansion is carried out at volume levels lower than the MTV. The Bayesian Optimal Phase II (BOP2) design is adopted, with each group expanded to 12 cases to evaluate the balance point between block success rate and motor function preservation.
  Interventions: Drug: Perform adductor canal block with liposomal bupivacaine.

INTERVENTIONS:
Drug: Perform adductor canal block with liposomal bupivacaine. — Patient Positioning: Supine with the surgical limb slightly flexed and externally rotated.
  Operator Setup: The operator stands on the surgical side, with the ultrasound machine positioned contralaterally. The anterior thigh is sterilized and draped.
  Ultrasound Technique: A high-frequency (5-12 MHz) linear ultrasound probe (Sonosite M-Turbo), protected by a 3M Tegaderm dressing, is placed perpendicular to the skin at the midpoint between the femoral trochanter and the superior patellar margin. The probe is maneuvered to visualize the adductor canal structures.
  Needle Insertion: After local anesthesia at the insertion site, a 22G 80 mm needle is advanced using an in-plane technique until the tip reaches the triangular hypoechoic area lateral to the femoral artery. Following negative aspiration for blood, 1.33% liposomal bupivacaine is injected around the target site.

SUMMARY:
Building on Bayesian design methodologies from volume optimization studies of ropivacaine in shoulder surgery, this study pioneers the application of a seamless dose-finding strategy in knee ACB. Utilizing advanced statistical models (BOIN/BOP2 design), we aim to systematically evaluate the volume-effect relationship of liposomal bupivacaine, providing precise dosing recommendations to advance personalized and optimized analgesic protocols for knee surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective general anesthesia for unilateral knee joint surgery.
* Patients who provide informed consent.
* Aged between 18 and 65 years old, regardless of gender.
* American Society of Anesthesiologists (ASA) physical status classification of Ⅰ to Ⅲ
* Body mass index (BMI) ≤ 35 kg/m².

Exclusion Criteria:

* Femoral neuropathy.
* Coagulation dysfunction.
* Allergy to local anesthetics.
* Infection at the puncture site.
* History of chronic pain or opioid use.
* Pregnancy.
* Diabetes mellitus and peripheral neuropathy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of the decline in the motor function of the quadriceps femoris muscle | Before block and 30 minutes after block
  The maximum voluntary isometric contraction (MVIC) of the quadriceps femoris muscle is measured using a handheld dynamometer (HHD) and then re - measured 30 minutes after the block. A decrease in muscle strength of ≥ 25% is defined as a significant impact on motor function.
The success rate of the block | 30 minutes after block
  Sensory block at 30 minutes after surgery (pinprick test at several sites in the area innervated by the saphenous nerve) and a resting NRS score ≤ 3 points. The sensory block is evaluated using a pinprick test for sensation. This test is performed before the adductor canal block (baseline) and every 5 minutes after the nerve block until 30 minutes have elapsed or the surgery begins. The sensory test is carried out in the distribution area of the saphenous nerve (medial side of the lower leg), as well as on the anterior, medial, lateral, and posteromedial sides of the surgical knee joint, and above the patella. A sensory score of 2 indicates normal sensation, 1 indicates hypoesthesia, and 0 indicates no sensation. We define a successful adductor canal block as the occurrence of sensory block in the surgical knee joint within 30 minutes after the nerve block, that is, the loss of sensation to the pinprick (sensory score of 1 or lower).

SECONDARY OUTCOMES:
Numerical Rating Scale scores during resting/movement | At 30 minutes, 1 hour, 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours after surgery
  The NRS (Numeric Rating Scale) scores range from 0 to 10 in total. A score of 0 represents no pain, while a score of 10 indicates severe pain. A score of 0 to 3 indicates mild pain, which is tolerable and does not affect sleep. A score of 4 to 6 indicates moderate pain, which is more obvious and will somewhat interfere with the patient's daily life and sleep, but is still bearable. A score of 7 to 10 indicates severe pain, which is intense and difficult to endure, seriously affecting the patient's daily life and sleep. The lower the score, the better the analgesic effect of the adductor canal block performed with liposomal bupivacaine.
Consumption of opioid drugs | within 48 hours after surgery
  converted into morphine equivalent, mg. After performing the adductor canal block with liposomal bupivacaine, the lower the consumption of opioid drugs, the better the effect of nerve block and the more prolonged the blocking duration.
Duration of analgesia | within 48 hours after surgery
  The time from the completion of the block to the first need for rescue analgesia.
The time of the first out-of-bed activity | within 48 hours after surgery
  Observe the impact of adductor canal block on the patient's motor function. If the patient can get out of bed and move for the first time within a relatively short and reasonable period, it usually indicates that the nerve block has a good effect. It can effectively relieve pain without excessively affecting the patient's motor function, enabling the patient to regain a certain degree of activity ability at an earlier stage.
Patient satisfaction | within 48 hours after surgery
  Total score of 10 points (0 points: extremely dissatisfied, 10 points: extremely satisfied). Higher scores indicate greater patient satisfaction and better efficacy of nerve block.
Satisfaction with postoperative rehabilitation | before discharge
  The patient's self-evaluated recovery experience (Likert 5-point scale). The Likert five-point scale employs an odd-numbered grading system (5-point scale), with each item corresponding to five options representing an intensity gradient of attitudes or experiences. Common expressions include:
  Strongly Disagree / Very Poor (1 point) Disagree / Poor (2 points) Neutral / Average (3 points) Agree / Good (4 points) Strongly Agree / Very Good (5 points) The total score is calculated by summing the scores of all items, reflecting the overall positivity of the evaluated experience (e.g., recovery experience).
The decline range of the quadriceps femoris muscle strength | 30 minutes after block
  The percentage change in muscle strength 30 minutes after the block compared to the baseline level.
Toxic reactions of local anesthetics (such as tinnitus, convulsions) | 7 days after surgery
  Pay attention to avoiding blood vessels. Aspirating during drug injection can reduce the toxic reaction of local anesthetics caused by the entry of local anesthetics into the bloodstream.
Neurological complications(numbness, tingling pain, muscle weakness) | within 30 minutes after the completion of the block
  Observe whether there is nerve injury. Muscle Strength Grading Standards (0-5 Scale) Assessment Method: To assess for neurological complications, inquire whether the patient experiences pain and if numbness is present in the saphenous nerve distribution area.
  Assess muscle strength levels through resistance-based grading. Grade 0 : No muscle contraction (complete paralysis) Limbs show no movement or tension.
  Grade 1 : Slight muscle contraction without joint movement Muscle twitching visible, no limb motion.
  Grade 2: Joint movement possible horizontally but cannot resist gravity Leg slides on bed but cannot lift.
  Grade 3 : Can complete motions against gravity but cannot resist external resistance Lifts leg off the bed but collapses under light pressure.
  Grade 4: Can resist partial external force but weaker than normal Holds position against mild resistance but fatigues quickly.
  Grade 5: Normal strength, fully resists resistance.
Whether it affects the sciatic nerve | within 48 hours after surgery
  Examine whether the sensory and motor function of the sciatic nerve is impaired
Incidence of Falls | 7 days after surgery
  he incidence of falls can reflect the impact of nerve block on quadriceps muscle strength; a higher incidence indicates a greater effect on motor function.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Shi, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Chen CM, Yun AG, Fan T. Continuous Bupivacaine Infusion versus Liposomal Bupivacaine in Adductor Canal Block for Total Knee Arthroplasty. J Knee Surg. 2022 Sep;35(11):1268-1272. doi: 10.1055/s-0040-1722661. Epub 2021 Feb 15. PMID 33588474
- [Background] Wang C, Zhang Z, Ma W, Li H, du X. Locating Adductor Canal and Quantifying the Median Effective Volume of Ropivacaine for Adductor Canal Block by Ultrasound. J Coll Physicians Surg Pak. 2021 Oct;31(10):1143-1147. doi: 10.29271/jcpsp.2021.10.1143. PMID 34601831
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Abdallah FW, Mejia J, Prasad GA, Moga R, Chahal J, Theodoropulos J, Dwyer T, Brull R. Opioid- and Motor-sparing with Proximal, Mid-, and Distal Locations for Adductor Canal Block in Anterior Cruciate Ligament Reconstruction: A Randomized Clinical Trial. Anesthesiology. 2019 Sep;131(3):619-629. doi: 10.1097/ALN.0000000000002817. PMID 31246607